CLINICAL TRIAL: NCT01073046
Title: Naso-gastric/Jejunal Tube Placement After Sub-total Gastrectomy. A Multicenter Prospective Randomized Trial
Brief Title: Gastric Decompression After Sub-total Gastrectomy
Status: Completed | Type: Observational
Sponsor: Catholic University, Italy (Other)
Collaborators: Italian Research Group For Gastric Cancer - IRGGC (Unknown)
Responsible Party: Principal Investigator, Fausto Rosa, MD, Catholic University, Italy
Other Study IDs: 1053222
Record Dates: First submitted 2010-02-01; First posted 2010-02-23 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2010-01

CONDITIONS: Gastric Cancer
Keywords: Naso-Gastric/Jejunal Tube; Sub-total Gastrectomy; Gastric Cancer; Decompression; Discomfort; Complications
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Place Naso-Gastric/Jejunal Tube Group: In this group a silastic naso-gastric/jejunal tube is placed (Rusch® distributed by Teleflex Medical Srl)
  Interventions: Device: Naso-Gastric/Jejunal Tube
- No Naso-Gastric/Jejunal Tube Group: In this group a silastic naso-gastric/jejunal tube is not placed

INTERVENTIONS:
Device: Naso-Gastric/Jejunal Tube — Silastic Naso-Gastric/Jejunal Tube (Rusch® distributed by Teleflex Medical Srl)
  Other Names: Rusch® distributed by Teleflex Medical Srl
  Groups: Place Naso-Gastric/Jejunal Tube Group

SUMMARY:
The purpose of this study is to test the utility of the nasogastric tube, which is used to decompress and as "guardian" of gastro-jejunal anastomosis, in patients undergoing distal subtotal gastrectomy for gastric cancer with reconstruction according to Billroth II or according Roux.

DETAILED DESCRIPTION:
A silastic naso-gastric tube (Rusch® distributed by Teleflex Medical Srl) is used in the naso-gastric/jejunal tube group

ELIGIBILITY:
Inclusion Criteria:

* All people subjected to subtotal gastrectomy for distal gastric adenocarcinoma.

Exclusion Criteria:

* People undergoing enteral nutrition through naso-jejunal tube

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be included, using a randomization list provided to each center, in one of two groups:
  1. placement of a polyurethane nasogastric/jejunal tube, preferentially 12-14 Fr;
  2. no feeding tube placement.
Sampling Method: Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Influence of Naso-Gastric/Jejunal Tube on Postoperative complications | 2 years

SECONDARY OUTCOMES:
Influence of Naso-Gastric/Jejunal Tube on Postoperative Patient's Comfort | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Digestive Surgery, Catholic University, Rome, Italy

REFERENCES:
- [Derived] Pacelli F, Rosa F, Marrelli D, Morgagni P, Framarini M, Cristadoro L, Pedrazzani C, Casadei R, Cozzaglio L, Covino M, Donini A, Roviello F, de Manzoni G, Doglietto GB. Naso-gastric or naso-jejunal decompression after partial distal gastrectomy for gastric cancer. Final results of a multicenter prospective randomized trial. Gastric Cancer. 2014 Oct;17(4):725-32. doi: 10.1007/s10120-013-0319-x. Epub 2013 Nov 30. PMID 24292257